CLINICAL TRIAL: NCT03286660
Title: Chair Rise Tests for a Simplified Evaluation of Functional Response After a Rehabilitation Program in Patients COPD.
Brief Title: 3 Minutes Chair Rise Test (3CRT) in Patients With COPD
Acronym: 3CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Boehringer Ingelheim (Industry); HYLAB, Physiopathologie de l'exercice (Unknown)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013_58; 2014-A00856-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-09-09; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Evaluations; Rehabilitation; COPD
Keywords: Exercise tests; COPD; Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD patients (Other): All convenient COPD patients admitted in real life for a rehabilitation program were included.
  Exercises consist on a Chair Rise Tests and short questionnaire were added to the usual tools for the evaluation.
  Interventions: Diagnostic Test: Chair Rise Tests and short questionnaire

INTERVENTIONS:
Diagnostic Test: Chair Rise Tests and short questionnaire — Exercises consist on a Chair Rise Tests and short questionnaire It is a functional test evaluating the number of chair rise over a given time and / or frequency.
  This test is combined with a questionnaire to collect quantitative and qualitative information:
  * dyspnea and muscular fatigue at rest before the start of the test and at the end of the exercise
  * Saturation at rest, and at the end of the exercise
  * the number of total a chair rise

SUMMARY:
Improvement in the functional functioning and dyspnea of COPD patients after a rehabilitation program (RHB) is assessed by exercise tests and questionnaires difficult to replicate outside specialized centers.

In order to monitor the eventual decline of patients in the course of their RHB management, Chair Rise Tests (3CRT-1CRT-5STS) and short questionnaires were developed (CAT-DIRECT). The goal of this prospective, multicenter, real-life study is to compare the change in several functional function tests and questionnaires of quality of life and dyspnea related to daily activities. In addition, MCIDs of the 3CRT and the DIRECT questionnaire (Disability Related to COPS Tool) were specified.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COPD Gold II to IV
* Patient admitted for a rehabilitation program in real life
* Person affiliated to the Social Security or beneficiary of such a scheme
* Informed and written consent by patient or legal representative

Exclusion Criteria:

* Patient limited by reduced locomotor activity or joint pain that compromises their participation in a rehabilitation program
* Patients with a performance less than 250 meters during 6MWT
* Non-stable cardiac disease
* Any other lung disease than COPD
* Person subject to a legal protection measure

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

PRIMARY OUTCOMES:
Change of number of rise during 3 minutes Chair Rise Test (3CRT) | At Baseline, at 2 and 8 weeks.
  The change of total number of rise during a 3 minutes Chair Rise Test (3CRT) from baseline

SECONDARY OUTCOMES:
Change of number of rise during 1 minute Chair Rise Test (1CRT) | At Baseline, at 2 and 8 weeks.
  The change of total number of rise during a 1 minutes Chair Rise Test (3CRT) from baseline
Change of Time to perform 5 sit to stand | At Baseline, at 2 and 8 weeks.
  The change of Time to perform 5 sit to stand from baseline
The change of Total score for the DIsability RElated to COPD Tool (DIRECT) | At Baseline and at 8 weeks.
  Total Score
Difference in physiological response (SpO2 and HR) during the 3 Chair Rise Tests (3CRT-1CRT-5STS) | At Baseline, at 2 and 8 weeks.
  End SpO2 - End Heart Rate
Change in endurance time at constant power on cyclo ergometer, | At Baseline, at 2 and 8 weeks.
  The change of endurance time from baseline
Change of Voluntary Quadriceps force output | At Baseline, at 2 and 8 weeks.
  Change of Voluntary quadriceps force measurements (Mean of 3 maximal measurements) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bernard AGUILANIU, MD,PhD, Principal Investigator — University Grenoble Alps
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire, Grenoble
  - Hôpital Calmette, CHRU, Lille

REFERENCES:
- [Derived] Levesque J, Antoniadis A, Li PZ, Herengt F, Brosson C, Grosbois JM, Bernady A, Bender A, Favre M, Guerder A, Surpas P, Similowski T, Aguilaniu B. Minimal clinically important difference of 3-minute chair rise test and the DIRECT questionnaire after pulmonary rehabilitation in COPD patients. Int J Chron Obstruct Pulmon Dis. 2019 Jan 22;14:261-269. doi: 10.2147/COPD.S187567. eCollection 2019. PMID 30774324